CLINICAL TRIAL: NCT04270162
Title: New Intervention Protocol With Inspirometer to Improve Lung Capacity Versus Traditional Use of Inspirometer and the Effects of Respiratory Exercises in Hospitalized Patients: INSPUL-REHAB
Brief Title: New Intervention Protocol With Inspirometer Versus 2 Modalities of Pulmonary Intervention: INSPUL-REHAB
Acronym: INSPUL-REHAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Angeles Lomas (Other)
Responsible Party: Principal Investigator, Javier Eliecer Pereira Rodriguez, Project coordinator and Physiotherapist, specialist in cardiopulmonary rehabilitation, magister in health sciences, magister in palliative care and university professor., Hospital Angeles Lomas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JEPRodriguez
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breathing Exercises
Keywords: Inspiratory volume, expiratory volume, inspirometer.

STUDY DESIGN:
Intervention Model Description: Hospitalized patients who after the exclusion criteria will begin the investigation and organize into 3 groups. The present one will be distributed with a basic probabilistic sampling using a random number table, whose order will be randomized through the Microsoft Excel 16.0 program, being experimental group 1 (New intervention protocol with inspirometer), experimental group 2 (Use of inspirometer in a conventional way) and control group (breathing exercises without the use of inspirometer).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New intervention protocol with inspirometer (Experimental): Respiratory exercises without use of inspirometerwill be taken out 50% and 80% to have it as muscle strength training values for the respiratory muscles based on the contra-relax technique)
  Interventions: Device: Respiratory muscle training 1
- Protocol of use of inspirometer in a conventional way (Active Comparator): This gonna be a experimental group 2 with conventional use of the conventional way.
  Interventions: Other: Respiratory muscle training 2
- Respiratory exercises without use of inspirometer (Active Comparator): This group gonna be a control group with breathing exercises without the use of inspirometer.
  Interventions: Other: Respiratory muscle training 3

INTERVENTIONS:
Device: Respiratory muscle training 1 — For inspirometer, the participant sits and holds the device. Then put the mouthpiece of the inspirometer in the mouth. Be sure to make a good seal on the mouthpiece with your lips. And exhale (exhale) normally until you run out of air. And after that, inhale (inspire) slowly as much as possible. This maximum value will be taken as an indicative parameter of its maximum inspiratory capacity and 50 and 80% of that value will be determined so that the participant performs 1 set of 10 repetitions at 50% of their maximum value, 2 sets of 10 repetitions at 60% of its maximum capacity and ends with 1 series at 80% of its maximum capacity.
  It is highlighted that in each series before finishing and without stopping to rest, the participant must do 5 repetitions at 100% maximum capacity.
  In addition, the respiratory exercises that will be carried out by the 3 intervention groups.
  Other Names: Inspirometer 1
  Arms: New intervention protocol with inspirometer
Other: Respiratory muscle training 2 — Training of respiratory muscles under the protocol of conventional use. Which is that the participant sits and holds the device. Then put the mouthpiece of the inspirometer in the mouth. Be sure to make a good seal on the mouthpiece with your lips. And exhale (exhale) normally until you run out of air. And after that, inhale (inspire) slowly as much as possible. Repeat 10 times and use these indications for 3 sets.
  In addition, participants must perform different breathing exercises that are identical for the 3 intervention groups.
  Other Names: Inspirometer 2
  Arms: Protocol of use of inspirometer in a conventional way
Other: Respiratory muscle training 3 — The same exercises that apply to the participants of experimental group 1 and 2 will be performed. The only difference is that the participants of this group do not perform exercises with inspirometer.
  Other Names: Respiratory exercises without inspirometer
  Arms: Respiratory exercises without use of inspirometer

SUMMARY:
A clinical trial will be carried out in the area of physiotherapy and rehabilitation of the "Centro Integral de Rehabilitación S.C. at the Hospital Angeles Lomas" in Mexico. Which, will have 3 arms (1. New intervention protocol created by the main author in the use of the inspirometer, 2. Conventional use of the inspirometer, 3. breathing exercises without the use of inspirometer) with hospitalized patient population and whose purpose will be to determine the effectiveness of the new intervention protocol and compare it with the current protocol and respiratory exercises.

DETAILED DESCRIPTION:
A clinical trial will be carried out in the area of physiotherapy and rehabilitation of the "Centro Integral de Rehabilitación S.C. at the Hospital Angeles Lomas" in Mexico. Whose population will be hospitalized patients at the angeles lomas hospital. This research is carried out with the purpose of knowing and applying the technique of contra-relax at the muscular level but in this case extrapolated in the inspirometer. This project will have 3 arms (1. New intervention protocol created by the main author in the use of the inspirometer, 2. Conventional use of the inspirometer, 3. breathing exercises) with a population of hospitalized patients and whose purpose will be to determine the effectiveness of the new intervention protocol and compare it with the current protocol and respiratory exercises.

The present project will be carried out with hospitalized patients who meet the criteria of occlusion and who, after passing the exclusion criteria, become part of a randomized clinical trial type investigation with a basic probabilistic sampling through a random number table, which Your order will be random through the Microsoft Excel 16.0 program, so we will obtain an experimental group 1, which will be the new intervention protocol for the use of the inspirometer (The maximum inspiratory capacity will be obtained and that results will be taken out 50% and 80% to have it as muscle strength training values for the respiratory muscles based on the contra-relax technique), an experimental group 2 (Conventional use of the conventional way) and a control group (breathing exercises without the use of inspirometer).

After your hospital stay, the post-training changes of the different groups will be determined taking as a reference and control value the maximum inspiratory volume and the maximum expiratory volume. The variables to be determined will be: Fatigue, dyspnea, maximum inspiratory capacity, maximum expiratory volume, quality of life, vital signs (heart rate, respiratory rate, blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients cardiopulmonary pathologies
* Over 18 years of age
* Patients who sign informed consent
* Possibility of performing your training for 1 month
* Participants than will can to go everyday for intervention.
* Participants do not have any inconvenience when doing the questionnaires, tests and measures that the investigation demands.

Exclusion Criteria:

* Participants who had severe pain in the lower or upper limbs.
* Unstable angina.
* Heart rate >120 bpm (beats per minute) at rest.
* Systolic blood pressure >190 mmHg.
* Diastolic blood pressure >120 mmHg.
* Participants who had a positive contraindication make exercise were not admitted in the study.
* Participants to show hemodynamic instability without improving during any test or during the intervention process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory volume (ml) | 1 month of training
  It will be determined by using the inspirometer whose values are from 0ml to 5,000ml. This pre and post intervention value will be determined
Changes in the levels of Fatigue after intervention | 1 month of training
  Fatigue was assessed using the FACT-Fatigue Scale Scale (Fatigue Scale of the Functional Evaluation of Cancer Therapy), which is an inventory of 13 items that assesses the severity of cancer-associated fatigue (FAC) in the last week. with a scale of 0 to 4 and that with higher scores reflect a lower FAC.
Changes in the Dyspnoea a after intervention | 1 month of training
  Dyspnea is a respiratory difficulty that usually translates into shortness of breath. Dyspnea can be determined using the original Borg scale (Score from 0 to 20) or modified (Score from 0 to 10), in which the higher the number indicated by the participant, the higher the degree of dyspnea.
Changes in the levels of Quality of life after intervention: EORTC QLQ-C30 | 1 month of training
  For the quality of life, it is necessary to use the questionnaire called EORTC QLQ-C30 (Version 3), which has 30 questions, where each question will go with a score of 1 to 4 and the higher the final result the better the quality of life. participant's life.

SECONDARY OUTCOMES:
Pre and post intervention blood pressure (mmhg) | 1 month of training
  Blood pressure will be determined by using a baumanometer.
Pre and post intervention heart rate (number of beats per minute) | 1 month of training
  The heart rate will be determined by using a pulse oximeter and corroborated manually.
Pre and post intervention respiratory rate (breaths per minute) | 1 month of training
  Heart rate will be determined visually by the researcher.
Changes in the Body Mass Index after intervention (%): | 1 month of training
  it is a mathematical reason that associates the mass and the size of an individual. it is also known as the Quetelet index. This result is determined by the formula of weight/square size.
Changes in the Abdominal circumference after intervention (cm): | 1 month of training
  It is the measurement of the distance around the abdomen at a specific point. Abdominal circumference is used to diagnose and monitor abdominal obesity. The values are in centimeters and according to the population to be studied, the measurements must be less than 90cm for men and 80cm for women.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Integral de Rehabilitación S.C. en el Hospital Angeles Lomas, Estado de México, Huixquilucan, Mexico

IPD SHARING:
Plan to Share IPD: No
We don´t have any plan because The research will be carried out directly among the researchers of our center. However, it is highlighted that we will make our results available to other researchers so that they can carry out future research that supports our results and compares with other types of populations.